CLINICAL TRIAL: NCT02537730
Title: BIOCLEAN MPS (Multi-Purpose Solution) VII in Combination With Biofinity Lens: A Two Week Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVJ-EX-MKTG-1318
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bioclean MPS VII / comfilcon A combination (Active Comparator): Participants were randomized to the Bioclean MPS VII / comfilcon A combination for one week during the cross over study.
  Interventions: Device: Bioclean MPS VII; Device: comfilcon A
- Aosept Clearcare / comfilcon A combination (Active Comparator): Participants were randomized to the Aosept Clearcare / comfilcon A combination for one week during the cross over study.
  Interventions: Device: Aosept Clearcare; Device: comfilcon A

INTERVENTIONS:
Device: Bioclean MPS VII — PHMB (Polyhexamethylene biguanide) base Disinfecting and Cleaning system
  Arms: Bioclean MPS VII / comfilcon A combination
Device: Aosept Clearcare — Hydrogen Peroxide Disinfecting and Cleaning system
  Arms: Aosept Clearcare / comfilcon A combination
Device: comfilcon A — contact lens
  Other Names: Biofinity

SUMMARY:
Two week, Open Label, randomized, bilateral, crossover, 1 week of daily wear in each combination (lens / disinfecting cleaning system).

DETAILED DESCRIPTION:
To determine if patients are unreactive to the lens care solution / Biofinity combination. It is expected that there will be a total of three visits: V1 (Initial), V2 (1 week), & V3 (2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Is over 18 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Has a CL (contact lens) spherical prescription between -0.25D (Diopters) and -12.00D (inclusive)
* Has less than 1.00 D spectacle cylinder in each eye
* Is correctable to a visual acuity of 20/20 or better in both eyes
* Has clear corneas and no active ocular disease
* Has read, understood and signed the informed consent letter
* Is willing to comply with the wear schedule (at least 40hrs per week)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has never worn contact lenses before
* Currently wears rigid gas permeable contact lens
* Has a history of not achieving comfortable CL (contact lens) wear (5 days per week; > 8 hours per day)
* Has a CL prescription outside the range of -0.25D to -12.00D
* Has a spectacle cylinder greater than -0.75D of cylinder in either eye
* Has best corrected spectacle distant vision worse than 20/20 in ether eye
* Has any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has any ocular pathology or sever insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars
* Is aphakic
* Is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kodama, MD, PhD, Principal Investigator — Kodama Eye Clinic
Locations (3):
- Japan (3):
  - Kodama Eye Clinic, Joyo-shi, Kyoto
  - Higashihara Eye Clinic, Kameoka, Kyoto
  - Iwasaki Eye Clinic, Osaka, Osaka

RESULTS

PARTICIPANT FLOW:
Groups:
- Bioclean MPS VII Combo, Then Aosept Clearcare Combo: Participants were randomized to the Bioclean MPS (Multi-Purpose Solution) VII / comfilcon A combination for one week, then cross over to the alternative Aosept Clearcare / comfilcon A combination
  Bioclean MPS VII: PHMB (Polyhexamethylene biguanide) base Disinfecting and Cleaning system
  Aosept Clearcare: Hydrogen Peroxide Disinfecting and Cleaning system
  comfilcon A: contact lens
- Aosept Clearcare Combo, Then Bioclean MPS VII Combo: Participants were randomized to the Aosept Clearcare / comfilcon A combination for one week then cross over to the alternative Bioclean MPS (Multi-Purpose Solution) VII / comfilcon A combination.
  Aosept Clearcare: Hydrogen Peroxide Disinfecting and Cleaning system
  Bioclean MPS VII: PHMB (Polyhexamethylene biguanide) base Disinfecting and Cleaning system
  comfilcon A: contact lens
Period: First Intervention (7 Days)
Arm/Group | Bioclean MPS VII Combo, Then Aosept Clearcare Combo | Aosept Clearcare Combo, Then Bioclean MPS VII Combo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Bioclean MPS VII Combo, Then Aosept Clearcare Combo | Aosept Clearcare Combo, Then Bioclean MPS VII Combo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Participants were randomized to the Bioclean MPS VII / comfilcon A combination or Aosept Clearcare / comfilcon A combination for one week, then cross over to the alternative combination.
Arm/Group | Overall Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Ocular Health - Corneal Staining
Description: Corneal staining for Bioclean MPS (Multi-Purpose Solution) VII / comfilcon A combination and Aosept Clearcare / comfilcon A combination assessed by slit lamp. Grade 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bioclean MPS VII / Comfilcon A Combination | Aosept Clearcare / Comfilcon A Combination
Number analyzed (Participants) | 33 | 33
Number analyzed (Eyes) | 66 | 66
Eyes
  Normal | 45 | 53
  Trace | 21 | 13
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0

2. Secondary Outcome: Comfort
Description: Subjective ratings of comfort scores for Bioclean MPS VII / comfilcon A combination and Aosept Clearcare / comfilcon A combination were assessed at 1 week: after insertion, after 4 hours of wear, after 8 hours of wear, before removal, and after all day wear. Scale 0-10, 0=very bad/poor, 10=very good/excellent.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioclean MPS VII / Comfilcon A Combination | Aosept Clearcare / Comfilcon A Combination
Number analyzed (Participants) | 33 | 33
units on a scale
  After insertion | 9.24 (1.42) | 9.30 (1.54)
  After 4 hours of wear | 9.52 (0.71) | 9.44 (1.05)
  After 8 hours of wear | 8.99 (1.03) | 9.10 (1.16)
  Before removal | 8.55 (1.13) | 8.65 (1.39)
  All day comfort | 9.15 (0.85) | 8.89 (1.14)

3. Secondary Outcome: Dryness
Description: Subjective ratings of dryness for Bioclean MPS VII / comfilcon A combination and Aosept Clearcare / comfilcon A combination were assessed at 1 week: after insertion, after 4 hours of wear, after 8 hours of wear, before removal, and after all day wear. Scale 0-10, 0=very bad/poor, 10=very good/excellent.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioclean MPS VII / Comfilcon A Combination | Aosept Clearcare / Comfilcon A Combination
Number analyzed (Participants) | 33 | 33
units on a scale
  After Insertion | 9.67 (0.69) | 9.77 (0.65)
  After 4 hours of wear | 9.27 (0.87) | 9.38 (0.86)
  After 8 hours of wear | 8.65 (1.22) | 8.91 (1.03)
  Before removal | 8.26 (1.29) | 8.33 (1.35)
  All day dryness | 8.92 (1.00) | 8.92 (1.00)

4. Secondary Outcome: Stinging and Burning Sensation
Description: Subjective ratings of stinging and burning sensation for Bioclean MPS VII / comfilcon A combination and Aosept Clearcare / comfilcon A combination. Scale 0-10, 0=difficult to wear, 10=no sensation at all.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bioclean MPS VII / Comfilcon A Combination | Aosept Clearcare / Comfilcon A Combination
Number analyzed (Participants) | 33 | 33
units on a scale
  Stinging Sensation | 9.42 (0.93) | 9.50 (0.93)
  Burning Sensation | 9.97 (0.17) | 9.91 (0.38)

ADVERSE EVENTS:
Time Frame: From dispense up to two weeks for each study lenses
Arm/Group | Bioclean MPS VII / Comfilcon A Combination | Aosept Clearcare / Comfilcon A Combination
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other